CLINICAL TRIAL: NCT04752215
Title: A First-in-human Phase I, Non-randomized, Open-label, Multi-center Dose-escalation Trial of BI 765049 and BI 765049 + Ezabenlimab Administered by Parenteral Administration(s) in Patients With Malignant Solid Tumors Expressing B7-H6.
Brief Title: A Study Evaluating Different Doses of BI 765049 When Given Alone and When Given With Ezabenlimab to Patients With Advanced Solid Tumors Expressing the Protein B7-H6 on the Cell Surface
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1454-0001
Record Dates: First submitted 2021-02-11; First posted 2021-02-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Neoplasms, Carcinoma, Non-Small-Cell Lung, Pancreatic Neoplasms, Carcinoma, Hepatocellular, Head and Neck Neoplasms, Gastrointestinal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma; Pancreatic Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 765049 single treatment group (Experimental): BI 765049
  Interventions: Drug: BI 765049
- BI 765049 + ezabenlimab combination treatment group (Experimental): BI 765049 + ezabenlimab
  Interventions: Drug: BI 765049; Drug: ezabenlimab

INTERVENTIONS:
Drug: BI 765049 — BI 765049
Drug: ezabenlimab — ezabenlimab
  Arms: BI 765049 + ezabenlimab combination treatment group

SUMMARY:
This study is open to adults with advanced solid tumors whose previous cancer treatment was not successful. People can participate if their tumor has the B7-H6 marker or if they have colorectal cancer.

The study tests 2 medicines called BI 765049 and ezabenlimab (BI 754091). Both medicines may help the immune system fight cancer.

The purpose of this study is to find out the highest dose of BI 765049 alone and in combination with ezabenlimab the participants can tolerate. In this study, BI 765049 is given to people for the first time.

Participants can stay in the study for up to 3 years, if they benefit from treatment and can tolerate it. During this time, they get BI 765049 alone or in combination with ezabenlimab as infusion into a vein every 3 weeks.

The doctors check the health of the participants and note any health problems that could have been caused by BI 765049 or ezabenlimab. The doctors also regularly monitor the size of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated, written informed consent form (ICF) (ICF1 for B7-H6 testing for all patients except those with advanced or metastatic colorectal cancer (CRC); and ICF2 for all patients) describing the study in accordance with International Council on Harmonisation Good Clinical Practice (ICH-GCP) and local legislation prior to any trial-specific procedures, sampling, or analyses.
* Patient must be ≥18 years of age at the time of signature on the ICFs (ICF1 and ICF2).
* Patients with a histologically or cytologically confirmed diagnosis of an advanced, unresectable, and/or metastatic colorectal carcinoma (CRC), non-small cell lung cancer (NSCLC), hepatocellular carcinoma (HCC), head and neck squamous cell carcinoma (HNSCC), gastric carcinoma, and pancreatic carcinoma. At least 1 patient in each back-fill slot must be a non-CRC patient (i.e., NSCLC, HCC, HNSCC, gastric carcinoma, or pancreatic carcinoma).
* Patients with disease progression despite conventional treatment, intolerant to or not a candidate for conventional treatment, or with a tumor for which no conventional treatment exists.
* All patients must agree to the collection of tumor samples (as slides from archival diagnostic samples or fresh tumor biopsies) for confirmation of B7-H6 expression either at Screening visit 02 (for CRC patients) or Screening visit 01 (for all other patients). To qualify for a back-fill slot or recommended dose expansion (RDE) cohort, the patient must agree to the collection of mandatory pre-treatment and on-treatment fresh tumor biopsies.
* Patient diagnosed with advanced or metastatic CRC or patient with confirmed B7-H6 expression on tumor tissue sample (archived or fresh tumor biopsy) based on central pathology review.
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patient must have at least one evaluable target lesion outside of the central nervous system (CNS) as defined per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 separate from any lesion(s) identified for tumor biopsy. Tumor lesions that have been irradiated at least ≥28 days before the start of treatment, and have subsequently had documented progression, may be chosen as target lesions only in the absence of measurable lesions that have not been irradiated.
* Further inclusion criteria apply

Exclusion Criteria:

* Patient with a history of a major surgery within 28 days prior to first dose of BI 765049 (major according to the Investigator's and/or Medical Monitor's assessment).
* Patient with a history of a previous or concomitant malignancies. Patient with a malignancy considered effectively treated and cured by 'local treatment' within the last 2 years and that is distinct from the one treated in this trial will be allowed.
* Patient with known leptomeningeal disease or spinal cord compression due to disease.
* Patient requiring anticoagulant treatment which cannot be safely interrupted, if medically needed for a study procedure (e.g., biopsy) based on the opinion of the Investigator.
* History of systemic antimicrobials required for an infection within 7 days of first dose BI 765049.
* Patient with any of the following laboratory evidence of hepatitis virus infection. Test results obtained in routine diagnostics are acceptable for screening if done within 14 days before the ICF2 date:

  * Positive results of hepatitis B surface (HBs) antigen
  * Presence of hepatitis B core (HBc) antibody together with hepatitis B virus (HBV)-DNA
  * Presence of hepatitis C-RNA
* Patient with known human immunodeficiency virus (HIV) infection.
* Patient previous treatment history:

  * Treatment with a systemic anti-cancer therapy or investigational drug within 21 days or 5 half-lives (whichever is shorter) of the first administration of BI 765049.
  * Treatment with extensive field radiotherapy including whole brain irradiation within 14 days prior to first administration of BI 765049.
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) in any studied regimen | Up to 3 weeks
  defined as the highest dose with less than 25 percent (%) risk of the true dose limiting toxicity (DLT) rate being equal to or above 33 percent (%) during the MTD evaluation period
Number of patients with dose limiting toxicities (DLTs) in the maximum tolerated dose (MTD) evaluation period | Up to 3 weeks

SECONDARY OUTCOMES:
Maximum measured concentration of BI 765049 (Cmax) | Up to 36 months
Area under the concentration-time curve of BI 765049 over a uniform dosing interval τ (AUCτ) | Up to 36 months
Objective response based on Response Evaluation Criteria in Solid Tumors (RECIST v1.1) in patients with measurable disease | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of California Irvine, Orange, California
  - HealthONE, Denver, Colorado
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Florida Cancer Specialists-Sarasota-61670, Sarasota, Florida
  - Northwestern University, Chicago, Illinois
  - Norton Healthcare - Norton Cancer Institute - Louisville, Louisville, Kentucky
  - New York University Langone Medical Center, New York, New York
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tennessee Oncology, PLLC-Nashville-52568, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
- Princess Margaret Cancer Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com